CLINICAL TRIAL: NCT00976638
Title: Mastering Hospital Antibiotic Resistance, a Cluster Randomized Intervention Study in Intensive Care Units Throughout Europe (Work Package 3)
Brief Title: Clinical Trial to Reduce Antibiotic Resistance in European Intensive Cares
Acronym: MOSAR-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, MJM Bonten, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LSHP-CT-2007-037941; WP3
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Hospital Acquired Infections
Keywords: Antimicrobial Resistant Bacteria; Hospital acquired infections; Colonization; Bacteremia; MRSA; VRE; ESBL; Intensive Care; ICU
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chromogenic Arm (Active Comparator): Active surveillance of colonization with MRSA or VRE by chromogenic agar with isolation of positive patients.
  Interventions: Other: Chromogenic surveillance
- Molecular Arm (Active Comparator): Active surveillance of colonization with MRSA and VRE by PCR; and of ESBL by chromogenic agar with isolation of positive patients
  Interventions: Other: Molecular surveillance

INTERVENTIONS:
Other: Chromogenic surveillance — All admitted patients are screened on admission for MRSA and VRE by chromogenic agar and isolated when positive
  Other Names: chromogenic screening
  Arms: Chromogenic Arm
Other: Molecular surveillance — All patients are screened for MRSA and VRE by PCR; and for ESBL by chromogenic agar on admission. Positive patients are isolated
  Other Names: molecular screening
  Arms: Molecular Arm

SUMMARY:
Colonization of patients with Antimicrobial Resistant Bacteria (AMRB) like Methicillin Resistant Staphylococcus Aureus (MRSA), Vancomycin-Resistant Enterococcus (VRE) and Extended-Spectrum Beta-Lactamases (ESBL) enterobacteriaceae leads to infections; and ultimately to adverse outcomes (eg prolonged hospital stay, death). This is an urgent problem in Europe, especially in Intensive Care Units (ICUs).

In this trial, colonization of patients with these AMRB will be assessed in the baseline period (6m). In phase 2 the effect of a Hygiene Improvement Program, including Chlorhexidine body washings and a Hand Hygiene training program, will be assessed (6m). In phase 3 units will be randomized to either Active Surveillance with Chromagar based tests or a Molecular based tests.

Study Hypothesis: the abovementioned interventions will reduce ICU-acquired colonization rates with MRSA, VRE and ESBL.

DETAILED DESCRIPTION:
A cluster-randomized trial with a stepped wedge design will be conducted in adult ICU's throughout Europe

The MOSAR-ICU trial is motivated by three primary considerations:

1. Advances in behavioral sciences and research about (hand) hygiene compliance have allowed a better understanding of barriers to increase compliance with (hand) hygiene practices within healthcare institutions;
2. Recent investigations have identified new rapid tests, both chromogenic media and molecular based tests, which may help identifying previously unknown carriage of AMRB at the time of admission; and
3. Currently practiced procedures, such as regular surveillance of all patients and daily cleansing of ICU patients with Chlorhexidine, have not been evaluated properly for their effectiveness.

In conclusion, evidence base derived recommendations from prospective studies regarding the costeffectiveness of different control strategies are lacking.

This study assess the impact of the three interventions on ICU acquired colonisation rates for AMRB(MRSA,VRE and ESBL).

Study design: Multi-center, cluster-randomised clinical trial.

Study population: Adult patients admitted to the ICU.

Intervention: The first phase of the study will be a 6-month baseline period to determine acquisition rates of AMRB during current standard practice in the individual participating centers (including currently performed surveillance strategies). The second phase will consist of a Hygiene Improvement Program to improve standard precautions and hand hygiene; and daily washing of all ICU patients with Chlorhexidine gluconate (HIP; 6 months). In both periods Contact Precautions (contact isolation) will be implemented for carriers of AMRB, as identified upon clinical cultures and following current practice of individual wards. In the third phase of the study (12 months) units will be randomized, and all interventions of phase 2 will be continued in all units. Half of the units will implement surveillance (admission and twice weekly cultures) of all admitted patients for carriage of MRSA and VRE using chromogenic agar. The other half will add molecular based rapid testing of ALL admission cultures for MRSA and VRE in addition to twice weekly screening of all patients with Chromagar based tests for MRSA, VRE and ESBL.

Main study endpoints: ICU-acquired colonization rates with MRSA, VRE and ESBL.

Primary Objective: To evaluate the impact of enhanced standard barrier precautions and rapid screening with targeted isolation of patients carrying AMRB on transmission of AMRB.

Secondary Objectives:

* Evaluate the impact of interventions on ICU-acquired bacteremia rates with MRSA, VRE or ESBL.
* Evaluate the impact of the HIP intervention on frequency and quality of hand hygiene, the application of standard precautions and the use of contact precautions during patient care.
* Evaluate the effect of the three strategies on other patient outcomes, including length of stay and in hospital mortality.
* Evaluate the overall antibiotic use and effectiveness of empirical treatment of ICU-acquired bacteremia.
* Evaluate the effect of the three strategies on the incidence density of new acquisitions with MRSA, VRE and ESBL individually.

ELIGIBILITY:
Inclusion Criteria:

* colonization with either MRSA, VRE or ESBL is endemic
* at least one dedicated infection control physician
* ability to obtain, store and analyze surveillance cultures
* at least 8 ICU beds; all of which have possibility for mechanical ventilation
* ability to collect the data required for analysis
* written approval of the institution's IRB
* signed protocol signature page

Exclusion Criteria:

* burn units
* cardiothoracic units
* pediatric and neonatal ICUs
* ICU is currently using rapid diagnostic testing in their screening program for AMRB
* ICU is planning to enroll subjects in studies testing investigational agents for the purpose of eradicating or preventing colonization with MRSA, VRE or ESBL or devices or practice management strategies that have colonization and/or infection with AMRB as an outcome
* using SOD/ SDD or any topical antimicrobial therapy
* using chlorhexidine body washings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14318 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Colonization with MRSA, VRE and ESBL | On admission
  By taking surveillance swabs from nose, perineum and wounds (if present) on admission we will assess whether patients are colonized with MRSA, VRE and ESBL at the moment of ICU admission. Swabs will be processed on chromogenic agars.
Colonization with MRSA, VRE and ESBL | During ICU stay
  By taking surveillance swabs twice weekly from nose, perineum and wounds (if present) we will assess whether patients become colonized with MRSA, VRE and ESBL during ICU stay. Swabs will be processed on chromogenic agars.
  Note: for patients admitted for longer than 21 days, surveillance is reduced to once weekly.

SECONDARY OUTCOMES:
Incidence density of new acquisitions with MRSA, VRE and ESBL individually. | Acquired during ICU stay (median LOS 14 days)
  In phase 2, we implement a hygiene improvement program. We will assess if this program reduces the number of patients acquiring colonization with MRSA, VRE and ESBL. We will measure colonization as stated in the primary outcome measure.
  In phase 3, we will implement direct feedback of screening results, and isolation of colonized patients. Swabs will be processed either by chromogenic agar (a) or molecular tests (b). Thus, the effect of these interventions on incidence density of new acquisitions of MRSA, VRE or ESBL will be assessed.
ICU-acquired bacteremia rates with MRSA,VRE or ESBL. | Acquired during ICU stay (median LOS 14 days)
  We will collect data on all bacteremias occuring during ICU stay, after completion of the trial. We include all bacteremias with s aureus (MSSA and MRSA), e faecium/ e faecalis ("S" and "R") and enterobacteriaceae ("S" and "R"). Data will be collected from the microbiology labs.
28 day-mortality | 28 days
  We will collect length of stay, and disposition at d28 as well as disposition at discharge from the ICU. Data will be collected in the online CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, Prof, MD, Principal Investigator — UMC Utrecht
Locations (13):
- France (3):
  - Hopital Henri Mondor, Créteil
  - Raymond Poincare Hospital, Garches
  - Hopital Paris Saint Joseph, Paris
- Greece (2):
  - Laikon General Hospital, Athens
  - University General Hospital Attikon, Athens
- San Camillo Forlanini Hospital, Rome, Italy
- Paul Stradins University Hospital, Riga, Latvia
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Portugal (2):
  - Hospital Geral de Sto Antonio, Porto
  - Tras-os-Montes e Alto Douro, Vila Real
- Slovenia (2):
  - University Clinic of Respiratory and Allergic Diseases, Golnik
  - University Medical Center Ljubljana, Ljubljana
- Hospital Clinic Y Provencal, Barcelona, Spain

REFERENCES:
- [Derived] Derde LPG, Cooper BS, Goossens H, Malhotra-Kumar S, Willems RJL, Gniadkowski M, Hryniewicz W, Empel J, Dautzenberg MJD, Annane D, Aragao I, Chalfine A, Dumpis U, Esteves F, Giamarellou H, Muzlovic I, Nardi G, Petrikkos GL, Tomic V, Marti AT, Stammet P, Brun-Buisson C, Bonten MJM; MOSAR WP3 Study Team. Interventions to reduce colonisation and transmission of antimicrobial-resistant bacteria in intensive care units: an interrupted time series study and cluster randomised trial. Lancet Infect Dis. 2014 Jan;14(1):31-39. doi: 10.1016/S1473-3099(13)70295-0. Epub 2013 Oct 23. PMID 24161233